CLINICAL TRIAL: NCT00172536
Title: Effects of Exercise Training on Left Ventricular Function in Type 2 Diabetic Patients Post Coronary Artery Bypass Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Ying-Tai Wu, School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 9361701147
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Coronary Arteriosclerosis; Post Coronary Artery Bypass Grafting
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Other): Received oral general education about proper diet, regular physcial activity and other medical care if necessary
  Interventions: Other: Control
- Exercise training (Experimental): Received a supervised structure treadmill training
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Subjects attended a supervised treadmill training session three times per week in an outpatient facility for three months. Training duration was 30 minutes per session, including a 5-minute warm-up and cool-down phase. Training intensity was initially set at about 60% of HR reserve and close to the anerobic threshold (AT) and the gradually increased as tolerated.
  Arms: Exercise training
Other: Control — Subjects received general education including proper diet, regular physical activity or medical care if necessary through an interview with a physical therapist.
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the changes of cardiorespiratory fitness and left ventricular function in type 2 diabetes after uncomplicated coronary artery bypass graft (CABG) surgery.

We hypothesize that exercise capacity, left ventricular diastolic function, and biochemical data improves after 12-wk exercise training in patients with type 2 diabetes underwent CABG.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus have higher incidence of coronary artery disease or left ventricular dysfunction, particularly diastolic dysfunction. Coronary artery bypass surgery is known to decrease the mortality rate in diabetes. Further exercise training can improve their cardiorespiratory fitness and the control of risk factors in these patients. However, the extent of improvement and the mechanism, especially the changes in left ventricular function, in diabetes after exercise training have not been fully explored.

Subjects will be assigned to the intervention or control group by randomization. Subjects in the intervention group will receive 60% VO2 max moderate aerobic exercise training, twice per week under supervision and three times per week at home, for 12 weeks. All subjects receive left ventricular function test by echocardiography and impedance cardiography, graded maximal exercise test, and biochemical analyses of sugar and lipid before and after 12 weeks. Their dietary intake and physical activity will be inquired every 4 weeks by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* well-controlled diabetes
* no history of myocardial infarction
* stable post CABG for at least 3 months

Exclusion Criteria:

* heart failure
* valvular disease
* abnormal kidney or liver function
* cerebrovascular disease
* primary pulmonary disease
* other systemic or acute illness that may impede the testing or training

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-10; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | Three months after the start of the intervention
  Exercise capacity was assessed by peak oxygen uptake (VO2peak)via exercise testing. VO2peak was measured by a metabolic measurement system (Vmax229 Metabolic Measurement System, Sensor Medics, Anaheim, CA).
Diastolic heart function | Three months after the start of the intervention
  Echocardiographic examination including color B mode TDI with a commercially available 2.5- to 3.75-MHz phased array transducer (Philips, SONOS 5500, Andover, MA)was used to evaluate diastolic function.

SECONDARY OUTCOMES:
Endothelial function | Three months after the start of the intervention
  Examined by flow-mediated vasodilation
Hemodynamics | Three times after the start of the intervention
  Heart rate (HR) and stroke volume (SV) were collected at rest, during the exercise test, and during the recovery phase by a noninvasive bioimpedance cardiograph device (PhysioFlow PF-05, Manatec Biomedical, Paris, France). Cardiac output (CO) and arteriovenous oxygen difference ((a-v)O2 difference) were then determined by the following equations: CO=HR*SV and (a-v)O2 difference=VO2/SV*HR
Blood test | Three months after the start of the intervention
  Including fasting glucose, HbA1c, total cholesterol (TC), high-density liporpotein (HDL-c) and triglyceride (TG).

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Doctor, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan